CLINICAL TRIAL: NCT04437706
Title: Network-Targeted Strategies for Efficient Community SARS-CoV-2 (COVID-19) Sampling
Acronym: Snowball
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105430
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; SARS-CoV 2
Keywords: network analysis; contact tracing; respondent driven sampling
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and pharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants completing COVID-19 testing

SUMMARY:
The primary objective is to use "network targeted sampling design" to detect active and/or undiagnosed cases of COVID-19 in the community and determine the spread or distribution of 1) active infection, and 2) past exposure. The hypothesis is that there are many undiagnosed and/or asymptomatic people in the community who may be unknowingly spreading the virus or have been exposed and have antibodies. We propose to implement respondent-driven sampling (RDS) which leverages effort on the part of seed or index cases to recruit contacts for participation.

DETAILED DESCRIPTION:
Purpose and objective: The purpose of this study is to use community sampling to detect active, undiagnosed COVID-19 cases and/or determine the spread or distribution of active infection. The objective is to use a network targeted sampling design to direct testing to yield a higher proportion of results which indicate active infection and possibly differentiating between venues or communities where transmission is active and undiagnosed.

Study activities: A person who tests positive for COVID-19 will be given a set of "tokens" to give to contacts that will entitle these contacts to make an appointment to receive a test for COVID-19.

Population groups: The population group will include people with index cases of COVID-19 and their contacts for the past 14 days. As these contacts are tested and receive positive results, they will be given tokens to hand out to their contacts over the past 14 days. The network of positive cases will "blossom" to reveal community transmission and asymptomatic cases, thus giving researchers an indication of disease prevalence.

Data analysis: At the completion of each epoch and at the end of the study, we will scale the social networks up and conduct network analysis using SAS and the igraph package in R. These analyses will be applied in an ongoing manner to guide selection of seeds in subsequent epochs to ensure representativeness and to guide selection of alters to encourage longer referral chain lengths.

Risk/safety issues: The primary risks include discomfort from the nasal swab and risks from the venous blood draw used in testing and the potential loss of confidentiality. All efforts will be made to securely manage the data to ensure participant confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 test result -or- receipt of a coupon from a previous study participant
* Resident of Durham County (for seed participant only)
* Willing to undergo COVID-19 test nasopharyngeal swab for RT-PCR testing and blood draw for COVID-19 antibody testing
* Age 18+
* Speak and understand English

Exclusion Criteria:

* Currently receiving inpatient treatment for COVID-19
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (18+ years) in the community who have tested positive for COVID-19 or have been in close contact with someone who is known to be COVID-19 positive
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Active Infection | 12 months
  Number of participants with active COVID-19 infection
Number of Participants with Antibodies Indicating Past Exposure | 12 months
  Number of participants with antibodies indicating past exposure to SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Dana Pasquale, PhD, Principal Investigator — Duke University
Locations (1):
- Margaret Pendzich, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pasquale DK, Welsh W, Olson A, Yacoub M, Moody J, Barajas Gomez BA, Bentley-Edwards KL, McCall J, Solis-Guzman ML, Dunn JP, Woods CW, Petzold EA, Bowie AC, Singh K, Huang ES. Scalable Strategies to Increase Efficiency and Augment Public Health Activities During Epidemic Peaks. J Public Health Manag Pract. 2023 Nov-Dec 01;29(6):863-873. doi: 10.1097/PHH.0000000000001780. Epub 2023 Jun 28. PMID 37379511
- [Result] Pasquale DK, Welsh W, Bentley-Edwards KL, Olson A, Wellons MC, Moody J. Homophily and social mixing in a small community: Implications for infectious disease transmission. PLoS One. 2024 May 28;19(5):e0303677. doi: 10.1371/journal.pone.0303677. eCollection 2024. PMID 38805519

DOCUMENTS (1):
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04437706/ICF_000.pdf